CLINICAL TRIAL: NCT00635102
Title: Glycine and Oral D-Cycloserine in Alcoholic Patients and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 12449; VA Merit Grant (Other Grant/Funding Number: VA Merit Grant)
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence, Alcoholism, Glycine, D-Cycloserine
MeSH Terms: conditions — Alcoholism | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol dependent (Active Comparator): Alcohol dependent patients will receive 4 interventions
  Interventions: Drug: D-Cycloserine PO and Glycine IV; Drug: Placebo D-Cycloserine PO and placebo Glycine IV; Drug: Placebo D-Cycloserine PO and Glycine IV; Drug: D-Cycloserine PO and placebo Glycine IV
- Healthy subjects (Active Comparator): Healthy subjects will receive 4 interventions
  Interventions: Drug: D-Cycloserine PO and Glycine IV; Drug: Placebo D-Cycloserine PO and placebo Glycine IV; Drug: Placebo D-Cycloserine PO and Glycine IV; Drug: D-Cycloserine PO and placebo Glycine IV

INTERVENTIONS:
Drug: D-Cycloserine PO and Glycine IV — Test days will involve administration of D-Cycloserine in the morning in pill form then 4 hours later a 30 minute infusion of Glycine.
  Other Names: Glycine infusion; Cycloserine
Drug: Placebo D-Cycloserine PO and placebo Glycine IV — Placebo
  Other Names: placebo
Drug: Placebo D-Cycloserine PO and Glycine IV
Drug: D-Cycloserine PO and placebo Glycine IV

SUMMARY:
Question #1: Will glycine ameliorate cognitive deficits? Hypothesis #1: Based on positive findings conducted with glycine and milacemide, a glycine prodrug, in schizophrenia and dementia, we expect that glycine will ameliorate cognitive deficits.

Question #2: Will alcoholic patients show enhanced endocrinal effects to glycine? Hypothesis #2: Based on the dose-related effects of glycine in healthy subjects, we expect that glycine will increase the endocrinal response to glycine in alcoholic patients with, supposedly, dysregulated NMDA receptor function.

Question #3: Will D-cycloserine have ethanol-like effects? Hypothesis #3: If inhibition of NMDA receptor function is fundamental to the subjective effects of ethanol, then the NMDA antagonist properties of D-cycloserine should be recognized as ethanol-like (relative to placebo) in recently detoxified alcoholics and healthy subjects.

Question #4: Will D-cycloserine reverse cognitive benefits of glycine? Hypothesis 4: Based on the dose related NMDA antagonist activity of D-cycloserine, we expect that D-cycloserine will compete with the agonist activity of glycine and therefore it will reverse the cognitive benefits of glycine.

Question #5: Will D-cycloserine inhibit endocrinal effects of glycine? Hypothesis #5: If the agonist activity of glycine is necessary to determine endocrine response, then the dose-related NMDA antagonist properties of D-cycloserine should block these effects.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the interaction between glycine and D-cycloserine in alcoholic patients and healthy subjects. Preclinical studies have shown that compounds acting at the glycine site of the N-methyl-D-aspartate (NMDA) receptor complex, such as glycine, may reverse the effects of ethanol on the NMDA receptor function (Rabe et al., 1990). The amino acid glycine is a co-agonist of the NMDA receptor complex (Kemp et al., 1993). It binds to the strychnine-insensitive site and positively modulates the NMDA receptor (Mc Donald et al., 1990). Physiologically, the glycine site is not saturated, and administration of glycine can potentiate NMDA receptor mediated responses. In contrast, D-cycloserine (Hood et al., 1989) is a partial-agonist at the glycine site of the NMDA receptor, with dose-dependent NMDA antagonist properties. The NMDA antagonist activity of D-cycloserine should produce ethanol like-effects that can be reversed by the agonist glycine. This study is intended to evaluate possible contributions of the glycine site to the reduction of cognitive deficits of alcoholism and complements the current work at VA Connecticut Healthcare System on the NMDA antagonists in alcoholic and healthy subjects.

ELIGIBILITY:
Inclusion / Exclusion Criteria Alcoholic subjects:

* Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 70 yrs.
* Meet Diagnostic and Statistical Manual (DSM) IV criteria for alcohol dependence by structured clinical interview
* Meet von Knorring criteria for early onset (type II) alcoholism
* Without other DSM IV Axis I diagnoses by Structured Clinical Interview (SCID).
* Without lifetime history of other substance abuse diagnosis by SCID (excluding tobacco) and urine toxicology screen negative for drug of abuse.
* Medically and neurologically healthy on the basis of history, physical examination, sequential multiple analysis-computer (SMAC-20), complete blood count (CBC) w/diff. and EKG. In light of the proximity to alcohol dependence, liver function test (LFT) elevations of twice normal will be accepted into the study.
* Patients with stable medical problems may be included in the study if their medications have not been adjusted in the month prior to participation and if these medications lack prominent central nervous system (CNS) effects.
* Absence of alcohol within the past 15 days.
* Patients must be free of medications utilized to facilitate detoxification (lorazepam, oxazepam) for at least 3 days prior to initiating testing.
* Patients must have no history of alcoholic hallucinosis.
* Patients must not be in acute alcohol withdrawal as evidence by a score no more than 2 for each item of the Clinical Institute Withdrawal Assessment Scale
* Patients taking ethionamide or isoniazid will be not be allowed to participate in the study.

Inclusion / Exclusion Criteria Healthy subjects:

* Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 70 yrs.
* Absence of a lifetime substance abuse diagnosis by the non-patient version of the SCID.
* Medically and neurologically healthy on the basis of history, physical examination, SMAC-20, CBC w/diff. and EKG. In light of the proximity to alcohol dependence, LFT elevations of twice normal will be accepted into the study.
* Absence of alcohol within the past 14 days
* Healthy subjects will be matched to the patient group for age, sex and educational level.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1997-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Krystal, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Result] Krystal JH, Petrakis IL, Limoncelli D, Nappi SK, Trevisan L, Pittman B, D'Souza DC, Suckow RF. Characterization of the interactive effects of glycine and D-cycloserine in men: further evidence for enhanced NMDA receptor function associated with human alcohol dependence. Neuropsychopharmacology. 2011 Feb;36(3):701-10. doi: 10.1038/npp.2010.203. Epub 2010 Dec 1. PMID 21124304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Alcoholic subjects were recruited from the Substance Abuse Treatment Program at VA Connecticut Healthcare Systems in West Haven, through advertisements in newspapers and postings in the community. Healthy subjects were recruited from the advertisements in newspapers and postings throughout the community.
Groups:
- Alcoholic Subjects: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 70 yrs. who meet Diagnostic and Statistical manual (DSM) IV criteria for alcohol dependence by structured clinical interview
- Healthy Subjects: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 70 yrs who have been absence of a lifetime substance abuse diagnosis by the non-patient version of the structured clinical interview (SCID).
Period: Overall Study
Arm/Group | Alcoholic Subjects | Healthy Subjects
Started | 27 | 30
Completed | 20 | 22
Not Completed | 7 | 8
Not completed — Withdrawal by Subject | 7 | 8

BASELINE CHARACTERISTICS:
Population: 57 individuals signed consent forms, of the 57 individuals 27 were alcohol dependent and 30 were healthy subjects. Of the alcohol dependent subjects 20 completed, 3 completed part of the study and 4 withdrew from the study. Of the healthy subjects, 22 completed, 4 completed part of the study and 4 withdrew from the study.
Groups:
- Alcoholic Subjects: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 70 yrs. who meet DSM IV criteria for alcohol dependence by structured clinical interview
- Healthy Subjects: Male or female (post-menopausal, surgically sterile, or negative pregnancy test at screening and agreement to utilize an established birth control during the testing period) between the age of 21 and 70 yrs who have been absence of a lifetime substance abuse diagnosis by the non-patient version of the SCID.
- Total: Total of all reporting groups
Arm/Group | Alcoholic Subjects | Healthy Subjects | Total
Number analyzed (Participants) | 27 | 30 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 30 | 57
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.5) | 31.9 (10) | 37.9 (.17)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 7 | 7
  Male | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  United States | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scales of Similarity to Alcohol - Baseline
Description: Visual Analog Scales of Similarity to Alcohol data using the Likert scale (0 Not at all similar to alcohol -7 Extremely similar to alcohol) evaluating the similarity of drug effects to alcohol
Time Frame: Baseline
Population: Visual Analog Scales of Similarity to Alcohol data using the Likert scale (0 Not at all similar to alcohol -7 Extremely similar to alcohol) evaluating the similarity of drug effects to alcohol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.18 (0.50) | 0.05 (0.21)
  Glycine / Placebo | 0.25 (1.12) | 0.04 (0.20)
  Placebo / Cycloserine | 0.10 (0.30) | 0.04 (0.20)
  Placebo / Placebo | 0.24 (0.54) | 0 (0)

2. Primary Outcome: Visual Analog Scales of Similarity to Alcohol 60 Minutes Prior to Glycine Infusion
Description: as for outcome 1
Time Frame: 60 minutes prior to Glycine infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.77 (1.77) | 1.41 (1.65)
  Glycine / Placebo | 0.65 (1.27) | 0.67 (1.63)
  Placebo / Cycloserine | 0.48 (0.87) | 1.17 (1.66)
  Placebo / Placebo | 0.43 (0.93) | .025 (0.61)

3. Primary Outcome: Visual Analog Scales of Similarity to Alcohol 30 Minutes
Description: as for outcome 1
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.57 (1.17) | 1.81 (1.89)
  Glycine / Placebo | 0.60 (1.14) | 0.71 (1.45)
  Placebo / Cycloserine | 1.05 (1.56) | 1.21 (2.13)
  Placebo / Placebo | 0.43 (0.98) | 0.13 (0.34)

4. Primary Outcome: Visual Analog Scales of Similarity to Alcohol 60 Minutes
Description: as for outcome 1
Time Frame: 60 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.67 (1.494) | 1.81 (1.72)
  Glycine / Placebo | 0.75 (1.52) | 0.70 (1.43)
  Placebo / Cycloserine | 0.81 (1.21) | 1.46 (2.17)
  Placebo / Placebo | 0.24 (0.54) | 0.13 (0.45)

5. Primary Outcome: Visual Analog Scales of Similarity to Alcohol 120 Minutes
Description: as for outcome 1
Time Frame: 120 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.43 (1.08) | 0.41 (1.14)
  Glycine / Placebo | 0.3 (0.98) | 0.09 (0.29)
  Placebo / Cycloserine | 0.57 (0.87) | 0.29 (0.62)
  Placebo / Placebo | 0.10 (0.30) | 0.33 (1.44)

6. Secondary Outcome: Number of Drinks Felt Consumed at 60 Minutes Prior to Glycine Infusion
Description: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 60 minutes prior to Glycine infusion
Population: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Measure: Mean (Standard Deviation); unit: drinks felt consumed
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
drinks felt consumed
  Glycine / Cycloserine | 0.50 (1.34) | 0.70 (1.40)
  Glycine / Placebo | 0.30 (0.73) | 0.25 (0.61)
  Placebo / Cycloserine | 0.24 (0.54) | 0.75 (1.03)
  Placebo / Placebo | 0.05 (0.22) | 0.22 (0.52)

7. Secondary Outcome: Number of Drinks Felt Consumed at 30 Minutes
Description: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 30 minutes
Population: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Measure: Mean (Standard Deviation); unit: Number of Drinks Felt Consumed
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
Number of Drinks Felt Consumed
  Glycine / Cycloserine | 0.38 (1.32) | 0.68 (1.00)
  Glycine / Placebo | 0.20 (0.62) | 0.13 (0.34)
  Placebo / Cycloserine | 0.38 (0.74) | 0.38 (1.10)
  Placebo / Placebo | 0.24 (0.77) | 0.04 (0.20)

8. Secondary Outcome: Number of Drinks Felt Consumed at 60 Minutes
Description: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 60 minutes
Population: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Measure: Mean (Standard Deviation); unit: Number of Drinks Felt Consumed
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
Number of Drinks Felt Consumed
  Glycine / Cycloserine | 0.05 (0.22) | 1.24 (1.73)
  Glycine / Placebo | 0.5 (1.1) | 0.4 (0.9)
  Placebo / Cycloserine | 0.86 (1.65) | 0.83 (1.47)
  Placebo / Placebo | 0.05 (0.22) | 0.2 (0.58)

9. Secondary Outcome: Number of Drinks Felt Consumed at 120 Minutes
Description: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Time Frame: 120 minutes
Population: The Number of Drinks Scale asks subjects to report on the number of alcoholic drinks they felt they had consumed.
Measure: Mean (Standard Deviation); unit: Number of Drinks Felt Consumed
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
Number of Drinks Felt Consumed
  Glycine / Cycloserine | 0 (0) | 0.13 (0.34)
  Glycine / Placebo | 0.1 (0.45) | 0.21 (0.83)
  Placebo / Cycloserine | 0.05 (0.22) | 0 (0)
  Placebo / Placebo | 0 (0) | 0.04 (0.2)

10. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Subscale Sedation - Baseline
Description: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Time Frame: Baseline
Population: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 3.41 (5.76) | 1.91 (3.19)
  Glycine / Placebo | 3.3 (6.51) | 2.75 (3.77)
  Placebo / Cycloserine | 3.57 (6.71) | 1.83 (3.38)
  Placebo / Placebo | 5 (9.2) | 1.88 (3.58)

11. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) - Subscale Sedation 60 Minutes Prior to Glycine Infusion
Description: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Time Frame: 60 minutes prior to Glycine infusion
Population: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.23 (10.32) | 7.39 (6.97)
  Glycine / Placebo | 6.6 (9.68) | 3.79 (4.72)
  Placebo / Cycloserine | 7.24 (11.05) | 6.25 (7.88)
  Placebo / Placebo | 4.57 (8.64) | 3.67 (5.37)

12. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Subscale Sedation - 30 Minutes
Description: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Time Frame: 30 minutes
Population: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 7.14 (12.01) | 10.05 (10.06)
  Glycine / Placebo | 5.8 (10.56) | 5.87 (7.95)
  Placebo / Cycloserine | 5.2 (8.45) | 7.04 (10.66)
  Placebo / Placebo | 4.62 (8.23) | 3.58 (4.83)

13. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Subscale Sedation - 60 Minutes
Description: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Time Frame: 60 minutes
Population: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 5.29 (8.49) | 9.64 (10.98)
  Glycine / Placebo | 5.65 (11.62) | 5.83 (8.87)
  Placebo / Cycloserine | 8.48 (11.96) | 8.54 (11.84)
  Placebo / Placebo | 4.14 (7.4) | 2.54 (4.92)

14. Secondary Outcome: Biphasic Alcohol Effects Scale (BAES) Subscale Sedation - 120 Minutes
Description: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Time Frame: 120 minutes
Population: Self-report rating scale used to measure the sedative effects (0 not at all sedated - 70 extremely sedated) of alcohol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 3.57 (7.02) | 4.13 (7.21)
  Glycine / Placebo | 4.35 (8.56) | 1.67 (3.31)
  Placebo / Cycloserine | 4 (7.36) | 3.04 (4.69)
  Placebo / Placebo | 3.71 (7.72) | 1.25 (2.82)

15. Secondary Outcome: Visual Analog Scales (VAS) - Baseline
Description: Visual Analog Scales (VAS): Self-report rating scale used to measure high (0 not at all - 7 extremely)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.32 (0.78) | 0.22 (0.85)
  Glycine / Placebo | 0.5 (1.4) | 0.22 (0.85)
  Placebo / Cycloserine | 0.76 (1.64) | 0.25 (0.90)
  Placebo / Placebo | 0.48 (0.98) | 0.25 (0.90)

16. Secondary Outcome: Visual Analog Scales (VAS) - 60 Minutes Prior to Glycine Infusion
Description: Visual Analog Scales (VAS): Self-report rating scale used to measure high (0 not at all - 7 extremely)
Time Frame: 60 minutes prior to Glycine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.64 (1.22) | 0.82 (1.44)
  Glycine / Placebo | 0.68 (1.20) | 0.33 (0.92)
  Placebo / Cycloserine | 0.48 (1.08) | 0.96 (1.64)
  Placebo / Placebo | 0.38 (0.97) | 0.61 (1.31)

17. Secondary Outcome: Visual Analog Scales (VAS) - 30 Minutes
Description: Visual Analog Scales (VAS): Self-report rating scale used to measure high (0 not at all - 7 extremely)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.48 (0.98) | 1.05 (1.73)
  Glycine / Placebo | 0.65 (1.09) | 0.30 (0.70)
  Placebo / Cycloserine | 0.48 (0.93) | 0.79 (1.56)
  Placebo / Placebo | 0.52 (1.03) | 0.25 (0.90)

18. Secondary Outcome: Visual Analog Scales (VAS) - 60 Minutes
Description: Visual Analog Scales (VAS): Self-report rating scale used to measure high (0 not at all - 7 extremely)
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.52 (1.37) | 0.91 (1.41)
  Glycine / Placebo | 0.8 (1.58) | 0.22 (0.67)
  Placebo / Cycloserine | 0.6 (0.99) | 0.71 (1.49)
  Placebo / Placebo | 0.19 (0.40) | 0.17 (0.82)

19. Secondary Outcome: Visual Analog Scales (VAS) - 120 Minutes
Description: Visual Analog Scales (VAS): Self-report rating scale used to measure high (0 not at all - 7 extremely)
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.8 (1.54) | 0.35 (1.11)
  Glycine / Placebo | 0.55 (1.05) | 0.21 (0.83)
  Placebo / Cycloserine | 0.76 (1.61) | 0.29 (0.91)
  Placebo / Placebo | 0.24 (0.54) | 0.25 (0.90)

20. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Desire to Drink- Baseline
Description: Alcohol Craving Scale (ACS) Subscale: Desire to drink: Self-report rating scale used to measure desire to drink alcohol (0 No desire to drink alcohol - 100 Definitely desire to drink alcohol)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 7.62 (12.21) | 3.04 (7.03)
  Glycine / Placebo | 9.5 (17.01) | 2.5 (7.37)
  Placebo / Cycloserine | 5 (8.02) | 1.67 (4.82)
  Placebo / Placebo | 7.62 (10.91) | 0 (0)

21. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Desire to Drink - 60 Minutes Prior to Glycine Infusion
Description: as for outcome 20
Time Frame: 60 minutes prior to Glycine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 7.27 (10.77) | 2.61 (7.52)
  Glycine / Placebo | 8.5 (14.24) | 1.67 (6.37)
  Placebo / Cycloserine | 6.67 (11.97) | 3.04 (8.76)
  Placebo / Placebo | 4.76 (8.14) | 1.25 (4.48)

22. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Desire to Drink: - 30 Minutes
Description: as for outcome 20
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 9.05 (19.21) | 1.82 (6.65)
  Glycine / Placebo | 9 (14.83) | 2.17 (7.36)
  Placebo / Cycloserine | 8 (13.99) | 2.5 (7.37)
  Placebo / Placebo | 5.71 (10.28) | 2.08 (6.58)

23. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Desire to Drink - 60 Minutes
Description: as for outcome 20
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.5 (11.37) | 1.82 (6.65)
  Glycine / Placebo | 9 (15.18) | 2.17 (7.36)
  Placebo / Cycloserine | 10.48 (16.88) | 1.67 (6.37)
  Placebo / Placebo | 5.71 (9.78) | 2.08 (5.88)

24. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Desire to Drink - 120 Minutes
Description: as for outcome 20
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.19 (10.71) | 1.30 (4.58)
  Glycine / Placebo | 8 (13.99) | 1.667 (4.82)
  Placebo / Cycloserine | 9.05 (14.8) | 2.08 (6.58)
  Placebo / Placebo | 5.24 (9.28) | 2.08 (6.58)

25. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Mood Improvement - Baseline
Description: Alcohol Craving Scale (ACS) Subscale: Mood improvement : Self-report rating scale used to measure expected alcohol-related mood improvement (0 Not at all - 100 Definitely)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.67 (11.55) | 1.74 (4.91)
  Glycine / Placebo | 10.5 (16.69) | 0.42 (2.04)
  Placebo / Cycloserine | 6.82 (12.87) | 0.42 (2.01)
  Placebo / Placebo | 8.10 (13.65) | 0 (0)

26. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Mood Improvement - 60 Minutes Prior to Glycine Infusion
Description: as for outcome 25
Time Frame: 60 minutes prior to Glycine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 7.73 (14.78) | 0.87 (2.88)
  Glycine / Placebo | 8 (11.97) | 0.83 (4.08)
  Placebo / Cycloserine | 7.62 (11.79) | 1.30 (4.58)
  Placebo / Placebo | 6.19 (10.71) | 0.42 (2.04)

27. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Mood Improvement - 30 Minutes
Description: as for outcome 25
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 11.43 (22.2) | 0.91 (4.26)
  Glycine / Placebo | 8 (12.81) | 0.87 (4.17)
  Placebo / Cycloserine | 10.5 (14.68) | 0.42 (2.04)
  Placebo / Placebo | 6.67 (10.17) | 0.42 (2.04)

28. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Mood Improvement - 60 Minutes
Description: as for outcome 25
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 5.5 (9.45) | 0.46 (2.13)
  Glycine / Placebo | 8.5 (13.87) | 0.87 (4.17)
  Placebo / Cycloserine | 8.1 (12.5) | 0.83 (2.82)
  Placebo / Placebo | 6.67 (11.97) | 0.83 (4.08)

29. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Mood Improvement - 120 Minutes
Description: as for outcome 25
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.19 (11.61) | 0.87 (2.88)
  Glycine / Placebo | 7 (11.74) | 0.83 (4.08)
  Placebo / Cycloserine | 8.57 (14.24) | 0.42 (2.04)
  Placebo / Placebo | 7.62 (14.11) | 0.42 (2.04)

30. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Discomfort - Baseline
Description: Alcohol Craving Scale (ACS) Subscale: Discomfort: Self-report rating scale - subscale reflecting expected alcohol-related relief from discomfort (0 Not at all - 100 Definitely)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 8.1 (15.04) | 2.61 (6.19)
  Glycine / Placebo | 12.5 (18.6) | 1.67 (5.65)
  Placebo / Cycloserine | 7.73 (13.78) | 0.42 (2.04)
  Placebo / Placebo | 8.10 (13.65) | 0.42 (2.04)

31. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Discomfort - 60 Minutes Prior to Glycine Infusion
Description: as for outcome 30
Time Frame: 60 minutes prior to Glycine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.36 (11.36) | 1.30 (4.58)
  Glycine / Placebo | 8.95 (13.29) | 1.25 (4.48)
  Placebo / Cycloserine | 7.14 (11.02) | 0.44 (2.09)
  Placebo / Placebo | 10.48 (15.65) | 0.42 (2.04)

32. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Discomfort - 30 Minutes
Description: as for outcome 30
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 12.38 (20.47) | 1.82 (5.89)
  Glycine / Placebo | 8.95 (13.29) | 1.74 (5.76)
  Placebo / Cycloserine | 9.5 (13.56) | 0.42 (2.04)
  Placebo / Placebo | 8.57 (11.95) | 0.42 (2.04)

33. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Discomfort - 60 Minutes
Description: as for outcome 30
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 6.5 (11.82) | 1.36 (4.68)
  Glycine / Placebo | 10.5 (16.70) | 1.74 (5.76)
  Placebo / Cycloserine | 9.05 (15.46) | 0.42 (2.04)
  Placebo / Placebo | 6.19 (10.71) | 0.83 (4.08)

34. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Discomfort - 120 Minutes
Description: as for outcome 30
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 8.57 (13.52) | 1.14 (4.91)
  Glycine / Placebo | 9.5 (15.38) | 1.67 (5.65)
  Placebo / Cycloserine | 9.05 (15.78) | 0.42 (2.04)
  Placebo / Placebo | 6.19 (11.17) | 0.83 (4.08)

35. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Reduced Control of Alcohol Use - Baseline
Description: Alcohol Craving Scale (ACS) Subscale: Self-report rating scale used to measure reduced control of alcohol (0 Not at all - 100 Definitely)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 29.05 (36.59) | 93.48 (21.24)
  Glycine / Placebo | 35.5 (40.32) | 94.58 (20.64)
  Placebo / Cycloserine | 42.27 (42.64) | 99.17 (4.08)
  Placebo / Placebo | 41.43 (40.29) | 98.75 (4.48)

36. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Reduced Control of Alcohol Use - 60 Minutes Prior to Glycine Infusion
Description: as for outcome 35
Time Frame: 60 minutes prior to Glycine infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 30.46 (37.48) | 98.26 (4.91)
  Glycine / Placebo | 40.5 (42.49) | 95 (20.64)
  Placebo / Cycloserine | 36.67 (41.51) | 99.13 (4.17)
  Placebo / Placebo | 42.86 (42.33) | 99.17 (4.08)

37. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Reduced Control of Alcohol Use - 30 Minutes
Description: as for outcome 35
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 32.86 (40.27) | 99.1 (4.26)
  Glycine / Placebo | 36 (40.18) | 98.70 (6.26)
  Placebo / Cycloserine | 36.5 (40.56) | 99.17 (4.08)
  Placebo / Placebo | 36.67 (37.59) | 99.17 (4.08)

38. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Reduced Control of Alcohol Use - 60 Minutes
Description: as for outcome 35
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 34 (42.23) | 99.1 (4.26)
  Glycine / Placebo | 39.5 (43.34) | 99.13 (4.17)
  Placebo / Cycloserine | 25.71 (35.3) | 99.17 (4.08)
  Placebo / Placebo | 37.14 (40.52) | 99.17 (4.08)

39. Secondary Outcome: Alcohol Craving Scale (ACS) Subscale: Reduced Control of Alcohol Use - 120 Minutes
Description: as for outcome 35
Time Frame: 120 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 34.29 (40.94) | 98.26 (4.91)
  Glycine / Placebo | 33.5 (42.83) | 99.17 (4.08)
  Placebo / Cycloserine | 30.48 (39.05) | 99.17 (4.08)
  Placebo / Placebo | 36.67 (40.17) | 99.17 (4.08)

40. Secondary Outcome: Continuous Performance Task (CPT) - Distractibility A-Prime - 30 Minutes
Description: gordon diagnostic system is a continuous performance task (CPT) to measure distractibility - (A-Prime score range 0 minimum - 1 maximum - the higher number the better the performance)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.93 (0.14) | 0.1 (0.01)
  Glycine / Placebo | 0.97 (0.05) | 0.1 (0.01)
  Placebo / Cycloserine | 0.90 (0.15) | 0.1 (0.01)
  Placebo / Placebo | 0.96 (0.05) | 0.1 (0.01)

41. Secondary Outcome: Continuous Performance Task (CPT) - Vigilance - A-Prime Score 30 Minutes
Description: gordon diagnostic system is a continuous performance task (CPT) to measure Vigilance - (A-Prime score range 0 minimum - 1 maximum - The higher number the better the performance)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 0.98 (0.03) | 0.1 (0.01)
  Glycine / Placebo | 0.1 (0.01) | 0.1 (0.02)
  Placebo / Cycloserine | 0.1 (0.02) | 0.1 (0.01)
  Placebo / Placebo | 0.99 (0.02) | 0.1 (0.00)

42. Secondary Outcome: Hopkins Verbal Learning Task - Immediate Recall - 60 Minutes - Trial 1
Description: Hopkins Verbal Learning Task (HVLT) - measures verbal memory and hippocampus function. (Three immediate recall trials) (0 No words recalled - 12 all words recalled)
Time Frame: 60 minutes - Trial 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 5.29 (1.93) | 7.09 (1.81)
  Glycine / Placebo | 6.05 (1.91) | 8.52 (1.95)
  Placebo / Cycloserine | 5.48 (1.12) | 7.75 (1.82)
  Placebo / Placebo | 5.95 (1.66) | 8.2 (1.56)

43. Secondary Outcome: Hopkins Verbal Learning Task - Immediate Recall - 60 Minutes - Trial 2
Description: as for outcome 42
Time Frame: 60 minutes - Trial 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 7.67 (2.08) | 10.09 (1.88)
  Glycine / Placebo | 8.45 (1.96) | 11.09 (1.20)
  Placebo / Cycloserine | 7.1 (1.67) | 10.5 (1.18)
  Placebo / Placebo | 8.67 (1.83) | 10.96 (1.37)

44. Secondary Outcome: Hopkins Verbal Learning Task - Immediate Recall - 60 Minutes - Trial 3
Description: as for outcome 42
Time Frame: 60 minutes - Trial 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 8 (2.47) | 10.57 (1.59)
  Glycine / Placebo | 9.2 (2.14) | 11.48 (0.85)
  Placebo / Cycloserine | 8.48 (2.02) | 11.17 (0.82)
  Placebo / Placebo | 9.24 (1.64) | 11.67 (0.76)

45. Secondary Outcome: Hopkins Verbal Learning Task - Delay Recall - 90 Minutes
Description: Hopkins Verbal Learning Task (HVLT) - measures verbal memory and hippocampus function. (delay recall - 30 minutes after Trials 1-3 were given) (0 No words recalled - 12 all words recalled)
Time Frame: 90 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alcoholic Subjects | Healthy Subjects
Number analyzed (Participants) | 20 | 22
units on a scale
  Glycine / Cycloserine | 5.1 (3.43) | 9.7 (2.44)
  Glycine / Placebo | 7.75 (2.4) | 10.87 (1.39)
  Placebo / Cycloserine | 6.29 (2.78) | 10.21 (1.74)
  Placebo / Placebo | 8.25 (2.43) | 11.38 (1.28)

ADVERSE EVENTS:
Arm/Group | Alcoholic Subjects | Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/30
Other Adverse Events (participants affected / at risk) | 0/27 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes